CLINICAL TRIAL: NCT00531596
Title: A PHASE IV, OPEN-LABEL STUDY OF THE ADHESION AND DERMAL TOLERABILITY OF EMSAM (SELEGILINE TRANSDERMAL SYSTEM) IN HEALTHY ADULT SUBJECTS OF TWO AGE GROUPS (18 - 64 YEARS, AND 65 YEARS AND OLDER)
Brief Title: Evaluation of Adhesion and Dermal Tolerability of EMSAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Somerset Pharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: S9303-P0602
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2007-09-19 (Estimated); Status verified 2007-09

CONDITIONS: Healthy
Keywords: Elderly; Non Elderly; Healthy Volunteers
MeSH Terms: interventions — Selegiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): EMSAM 6mg/24hr
  Interventions: Drug: EMSAM (Selegiline Transdermal System) 6mg/24Hr
- B (Active Comparator): EMSAM 9mg/24Hr
  Interventions: Drug: EMSAM (Selegiline Transdermal System) 9mg/24Hr
- C (Active Comparator): EMSAM 12mg/24Hr
  Interventions: Drug: EMSAM (Selegiline Transdermal System) 12mg/24hr

INTERVENTIONS:
Drug: EMSAM (Selegiline Transdermal System) 6mg/24Hr — EMSAM 6mg/24HR
  Arms: A
Drug: EMSAM (Selegiline Transdermal System) 9mg/24Hr — EMSAM 9mg/24Hr
  Arms: B
Drug: EMSAM (Selegiline Transdermal System) 12mg/24hr — EMSAM 12mg/24Hr
  Arms: C

SUMMARY:
Examine adhesive and dermal tolerability of EMSAm 6mg/24hr and 12mg/24hr in healthy elderly and non-elderly subjects.

DETAILED DESCRIPTION:
The primary objectives of this study are to examine the adhesion characteristics and dermal tolerability (irritation) of EMSAM in two populations consisting of non-elderly (18 - 64 years) and elderly (65 years and older) healthy volunteers. EMSAM will be dosed over the range of proposed sizes for marketing [(6mg/24hr), (9mg/24hr), and (12mg/24hr)]. Adhesion and tolerability (irritation) will be examined at three different application site areas (upper torso [includes chest and back], upper arm, and upper thigh).

The secondary objective is to examine if the adhesion characteristics and dermal tolerability (irritation) of EMSAM may be influenced by the secondary factors such as gender, race, physical activity, and bathing/showering practices.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study participation, subjects will meet the following criteria:

* Able and willing to provide written informed consent.
* Able and willing to follow a modified diet.
* 18 years of age and older.
* Male or female.
* If female and of childbearing potential, subject must have a negative pregnancy screen at baseline and may not be lactating. Females of childbearing potential must demonstrate use of an acceptable form of birth control, such as hormonal contraceptive, intrauterine device or barrier method (i.e. condom w/spermicide). NOTE: Abstinence and partner vasectomy are not acceptable methods of contraception.
* In general good health as ascertained by physical examination, supine and standing vital signs, laboratory test results, 12 lead ECG and medical history.

Exclusion Criteria:

Any of the following conditions will exclude subjects from eligibility for study participation:

* Subjects with a past or present condition that includes any of the following:

  1. In the opinion of the Investigator, any significant cardiovascular disease or disorder including myocardial infarction, cardiac arrhythmia, hypertension or recurrent episodes of orthostatic hypotension.
  2. Any skin abnormalities at or near designated patch application sites that might interfere with the conduct or interpretation of the study including the presence of moles, blemishes, excess hair, scars, tattoos, sunburn or other marks on the application sites that may obscure grading of the site(s).
  3. Any known hypersensitivity, or related hypersensitivity, to selegiline or to skin adhesives (i.e. surgical tape, etc.).
  4. Any significant immunological, pulmonary, hematologic, endocrine and/or metabolic disease or disorder or severe or acute medical illness, such as, metastatic cancer, brain tumors, decompensated cardiac, hepatic or renal failure.
  5. Neurological disorders including delirium, history of significant head trauma, movement disorders, dementia, multiple sclerosis or stroke.
  6. Any psychiatric disorders (except personality disorders) requiring treatment or therapy within the last three months.
  7. Any mood disorder including MDD which is current or relapsed over the past three years.
  8. Attention deficit hyperactivity disorder or attention deficit disorder.
  9. Any other condition, illness or disorder that in the opinion of the Investigator would place the subject at significant risk or any inability to follow the requirements of the study regarding maintaining scheduled visits or patch applications.
  10. Known substance abuse or addiction.
  11. Any significant allergy, especially involving dermal manifestations.
  12. History of sun hypersensitivity and photosensitive dermatoses.
* Recent or current treatment with systemic or topical drugs or medications which can interfere with skin responses (i.e. steroids, corticosteroids, antihistamines or anti-inflammatory agents). Daily regimens of low-dose aspirin is acceptable.
* Current or anticipated use of meperidine, tricyclic antidepressants, or selective serotonin reuptake inhibitors (i.e., fluoxetine [Prozac], etc) and other antidepressant medications (e.g., SNRI's, MAOI's, buproprion, etc).
* Use of any herbal or homeopathic remedies (excluding vitamins, fish oil, echinacea, glucosamine, chondroitin or calcium)within 14 days of study drug administration, during study conduct and 14 days after the completion of the study medication.
* Participation in a clinical investigation within 28 days prior to baseline.
* Current use of any agents listed as contraindicated (Section 10.3.1.3) or as listed in the approved label

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-04; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Adhesion characteristics and dermal tolerability (irritation) of EMSAM in two populations consisting of non-elderly (18 - 64 years) and elderly (65 years and older) healthy volunteers. | 21 Days

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Goodhead, Study Chair — Somerset Pharmaceuticals
Locations (2):
- United States (2):
  - Hill Top Research, Scottsdale, Arizona
  - Hill Top Research, St. Petersburg, Florida